CLINICAL TRIAL: NCT03140709
Title: Non-Invasive, Highly Specific Detection of Oxytocin in Biological Fluids
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Giner, Inc (Other); Aptagen, LLC (Unknown); Fraunhofer Center for Manufacturing Innovation (Unknown); Rose Biotech, LLC (Unknown)
Responsible Party: Principal Investigator, Brendan Carvalho, Chief, Division of Obstetric Anesthesia Department of Anesthesiology, Perioperative and Pain Medicine, Stanford University School of Medicine, Stanford University
Other Study IDs: 36843
Record Dates: First submitted 2016-05-15; First posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Oxytocin; Pregnancy
Keywords: Salivary; Oxytocin; Induction; Labor
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and blood samples will be obtained from study participants to monitor oxytocin levels. Observational study. Standard of care management. Oxytocin assays during normal clinical care.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Induced vaginal delivery: Saliva samples will be obtained both during induction and infusion, every 15 minutes after each change in dose. An estimated total of 5 saliva samples will be collected from each patient. Therefore, the last collection point (sample 5) will be during the oxytocin infusion after the 4th dose change. In addition, 2 blood samples will be collected from 5 patients - one baseline sample and another sample at same time as last saliva sample.
  Interventions: Drug: Oxytocin
- Cesarian delivery: A total of 3 saliva samples will be collected from each patient - one at baseline preoperative, one intrapartum at least 15 min after starting the standard 250 ml/h oxytocin infusion, and one postpartum in post-anesthesia care unit (PACU) at least 15 min after starting the standard 125 ml/h oxytocin infusion. Therefore, the last collection point (sample 3) will be during the oxytocin infusion in PACU. In addition, 1 blood sample will be collected from each patient in this cohort - at same time as last saliva sample.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Induction-Vaginal Delivery: Begin at 1mU/min IV infusion and increase by 2mU/30min q30min to a max of 30mU/min. Postpartum infusion adjusted to 2U/hr.
  Cesarian Delivery: 1U bolus via IV at delivery, followed by 7.5U/hr up to 30U/hour max depending on uterine tone. Postpartum infusion adjusted to 2U/hr
  Other Names: Pitocin

SUMMARY:
This study will aid in the development of a research instrument for rapid and highly sensitive detection of perinatal salivary oxytocin, by non-invasive means. There will be two study cohorts: Induction of labor cohort (20) and Cesarean delivery cohort (5) for a total of 25 participants.The standard clinical protocols for administering oxytocin to human subjects at Lucile Packard Children's Hospital will be followed. Oxytocin will be prescribed and dosed as per standard of care with no change due to study enrollment. The study will only involve sampling of saliva and blood.

The general hypothesis to be tested is that 1) the sensor will accurately report the levels of oxytocin in saliva samples as compared with standard reference methods and 2) the sensor yields rapid (<20 minutes) oxytocin results with minimal discomfort to subjects. Overall, this will allow to optimize the administration of oxytocin, and for a better understanding of the blood concentration and effects of oxytocin on mother and child.

DETAILED DESCRIPTION:
Oxytocin, a neuropeptide hormone, plays an important role in the dynamic function of the brain and a variety of complex social behaviors including affiliation, sexual behavior, social recognition, and aggression. Oxytocin is best known for its role to facilitate the birth process through induction of uterine smooth muscle contractions. Oxytocin is primarily used to induce labor, and contract the uterus after delivery. Oxytocin is considered the first line uterotonic to prevent and treat uterine atony and manage postpartum hemorrhage. Currently, there is no instrument that is capable of point-of-care oxytocin detection. A practical research tool to monitor peripheral levels of both endogenous and exogenous oxytocin is therefore needed to better understanding the pharmacokinetics and pharmacodynamics of oxytocin in the mother, fetus and newborn. A better understanding of drug concentration and effect may lead to optimal dosing and better management of induction of labor and/or uterine atony after delivery.

With increased research on the importance of oxytocin monitoring, a bedside oxytocin monitor is envisioned that would allow healthcare professionals to improve our pharmacokinetic/dynamic understanding of oxytocin and to monitor and adjust the dose of oxytocin administered during childbirth. Currently, there is no instrument that is capable of point-of-care oxytocin detection.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, pregnant woman (37-41 weeks)
* Scheduled for induction of labor (not already in active labor) or cesarean section
* Ages 18-45 years old
* ASA physical status 1 or 2
* Singleton pregnancy
* Able and willing to sign consent

Exclusion Criteria:

* Women with any significant medical or obstetric condition (such as gestational hypertension, diabetes,coagulopathy, and renal impairment)
* Morbid obesity (BMI greater than/equal to 40)
* In active labor upon arrival to L&D

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 25 generally healthy, pregnant adult women of all ethnicities, between the ages of 18 and 45, admitted for scheduled induction of labor or Cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Quantification of salivary oxytocin assay levels | 15 minutes after dose change
  Test novel aptamer-based electrochemical assay for the detection and quantification of salivary oxytocin

SECONDARY OUTCOMES:
Quantification of blood oxytocin levels | 15 minutes after dose change
  Standard of care detection protocol for oxytocin blood levels to compare sensitivity and specificity of aptamer-based electrochemical assay

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Carvalho, MBBCh MDCH, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dyer RA, Butwick AJ, Carvalho B. Oxytocin for labour and caesarean delivery: implications for the anaesthesiologist. Curr Opin Anaesthesiol. 2011 Jun;24(3):255-61. doi: 10.1097/ACO.0b013e328345331c. PMID 21415725
- [Background] Butwick AJ, Coleman L, Cohen SE, Riley ET, Carvalho B. Minimum effective bolus dose of oxytocin during elective Caesarean delivery. Br J Anaesth. 2010 Mar;104(3):338-43. doi: 10.1093/bja/aeq004. PMID 20150347